CLINICAL TRIAL: NCT05694442
Title: The Effect of Lipmatte K on Lip Hydration and Brightening
Brief Title: The Effect of Lipmatte K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UMRAMREC002-22
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Aesthetic; Cosmetic; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lipmatte K (Experimental): Participants will used Lipmatte K everyday for 4 weeks
  Interventions: Other: Lipmatte K

INTERVENTIONS:
Other: Lipmatte K — Lipmatte K contain ingredients that may hydrate and brighten the lip

SUMMARY:
This study is conducted to evaluate the safety and the effectiveness of Lipmatte K on lip hydration and brightening. The study duration is 4 weeks and the lip assessment will be carried out at baseline, week 2 and week 4.The main questions this study aims to answer are:

1. The hydration effect of the product on lip.
2. The brightening effect of the product on lip.
3. To observe any adverse effect occurrence with the usage of the product.

ELIGIBILITY:
Inclusion Criteria:

* Malaysia citizen
* Female (age 30-55 years old)
* Lip with mild-to-moderate dryness

Exclusion Criteria:

* Subjects who have history of performing lips-related treatments such as lip augmentation (filler, botox, laser)
* Heavy lips desquamation or chapped lip conditions

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in lip roughness from baseline and at week 2 and 4 after using Lipmatte K | Baseline, Week 2, Week 4
  Degree of lip roughness for each participant's will be determined by dermatologist based on score 0 to 2 (0= no desquamations, 1 = slight desquamations and 2 = heavy desquamations)
Change in lip wrinkles from baseline and at week 2 and 4 after using Lipmatte K | Baseline, Week 2, Week 4
  Degree of lip wrinkle for each participant's will be determined by dermatologist based on score 0- 2 (0 = no/almost no vertical wrinkles, 1 = no deep vertical wrinkles and 2 = many deep vertical wrinkles)
Visual assessment of the lip from baseline and at week 2 and 4 after using Lipmatte K | Baseline, Week 2, Week 4
  Image of the lip will be captured using digital camera (Nikon D5100) to observed the brightening effect of the lipmatte
Adverse effect after using Lipmatte K | Week 4
  Based on adverse effect occurrence on participants that occur during study period (4 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No